CLINICAL TRIAL: NCT02695342
Title: Pilot Study of a Tailored Home Balance Exercise Program for Reducing Falls in Older Adults With COPD
Brief Title: Home Balance Pilot for Fall Reduction in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: West Park Healthcare Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Labarge-20004484
Record Dates: First submitted 2016-02-22; First posted 2016-03-01 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Balance; Falls; Exercise; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home balance exercise program (Experimental): The home-based exercise program will be tailored to address the underlying balance deficits in COPD and individualized according to each participant's ability. Physiotherapists will teach the program in four home visits over the first 6 weeks of the study; in the event of an exacerbation, a fifth visit will be provided to modify the program. Participants will be given an exercise DVD (with portable player), and will be instructed to perform the program 3 times/week for 6 months. Therapists will provide bi-monthly telephone support.
  Interventions: Behavioral: Home balance exercise program

INTERVENTIONS:
Behavioral: Home balance exercise program

SUMMARY:
There is a growing body of evidence demonstrating that older adults with COPD have important problems with their balance and a high incidence of falls compared to those of a similar age. This research will explore the feasibility and preliminary effects of a tailored 6-month home balance exercise program for reducing falls in older adults with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is highly prevalent among older adults and is a leading cause of death, disability and hospitalization in Canada. There is a growing body of evidence demonstrating that older adults with COPD have important problems with their balance and a high incidence of falls compared to those of a similar age. This research will explore the feasibility and preliminary efficacy of a tailored 6-month home balance exercise program for reducing falls in older adults with COPD.

The primary objective of this pilot study is to determine the feasibility of a tailored home balance intervention for older adults with COPD in terms of recruitment, retention and adherence. The secondary objective is to examine the within-subject effects of the home-balance intervention on intermediate outcomes linked to falls including balance, functional strength and self-reported disability.

Thirty-five older adults with COPD will be recruited from respirology clinics at West Park Healthcare Centre (Toronto) and the Firestone Institute for Respiratory Health (Hamilton) to participate in a single-group, non-randomized clinical trial. Eligible participants will be enrolled in a 6-month balance home exercise intervention. The home program will be supervised by a physiotherapist and outcome measures will be collected at home at baseline, 3- and 6-months by a research assistant not involved in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of COPD;
* age ≥ 60 yrs;
* a history of 1 or more falls in the previous year;
* ability to provide written informed consent.

Exclusion Criteria:

* inability to communicate in English;
* history of significant cardiovascular disease;
* marked decrease in arterial oxygen saturation at rest or during previous assessments of exercise capacity;
* severe cognitive impairment;
* evidence of a condition that severely limits mobility and may jeopardize safety;
* completion of a course of rehabilitation in the last 6 months or on a wait list for admission to rehabilitation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-01; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Percentage of eligible patients that consent to enroll in the study
Retention rate | 6 months
  Percentage of the sample that complete all 3 outcome assessments
Compliance | 6 months
  Mean number of prescribed exercise sessions completed

SECONDARY OUTCOMES:
Berg Balance Scale | baseline, 3 months, 6 months
  Measure of balance
Balance Evaluation Systems Test (BESTest) | baseline, 3 months, 6 months
  Measure of balance
Activity-Specific Balance Confidence questionnaire | baseline, 3 months, 6 months
  Measure of balance confidence
30-second Sit-to-Stand Test | baseline 3 months, 6 months
  Measure of functional lower body strength
Self-reported function (PF-10) | baseline, 3 months, 6 months
  Physical function sub-scale of the Medical Outcomes Study 36-item Short-form Health Survey

OTHER OUTCOMES:
Number of falls reported per participant | Baseline, 6 months
  Fall history will be measured at baseline and prospectively using monthly fall diaries
Patient satisfaction questionnaire | 6 months
  Measure of patient satisfaction
Adverse events | 6 months
  Adverse event history will be tracked

CONTACTS AND LOCATIONS:
Overall Officials: Marla K Beauchamp, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Firestone Institute for Respiratory Health, St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - West Park Healthcare Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No